CLINICAL TRIAL: NCT06199973
Title: Injection of SHR-A1811 Versus Physician Choiced Treatment in Patients With Advanced Colorectal Cancer Who Had Failed to Respond to Oxaliplatin, 5-fu, and Irinotecan
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-309
Record Dates: First submitted 2023-12-26; First posted 2024-01-10 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Advanced Colorectal Cancer
MeSH Terms: interventions — trifluridine tipiracil drug combination; regorafenib; HMPL-013

STUDY DESIGN:
Intervention Model Description: SHR-A1811 for Injection with TAS-102
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR-A1811 (Experimental)
  Interventions: Drug: SHR-A1811
- physician choiced treatment (Experimental): include: TAS-102, or Regorafenib, or Fruquintinib
  Interventions: Drug: TAS-102, Regorafenib , Fruquintinib

INTERVENTIONS:
Drug: SHR-A1811 — SHR-A1811(4.8 mg/kg) was administered intravenously on the first day of each cycle, once every 3 weeks (Q3W)
  Arms: SHR-A1811
Drug: TAS-102, Regorafenib , Fruquintinib — physician choiced treatment,include: TAS-102(35 mg/m2, maximum 80 mg per dose), twice daily (BID) , once every 4 weeks (Q4W) , up to 3 years; or Regorafenib 160mg, once daily (QD) , once every 4 weeks (Q4W) , up to 3 years; or Fruquintinib 5mg once daily (QD) , once every 4 weeks (Q4W) , up to 3 years.
  Arms: physician choiced treatment

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of SHR-A1811 in advanced colorectal cancer subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Unresectable locally advanced or distant metastatic RAS/RAF wild-type colorectal cancer diagnosed histologically or cytologically;
2. After treatment with oxaliplatin, 5-fluorouracil (such as 5-FU, Capecitabine) , irinotecan (DMMR/MSI-H subjects also need anti-PD-1/PD-L1 antibody treatment failure) ;
3. According to the response evaluation criteria for solid tumors (RECIST 1.1) , having at least one measurable lesion, measurable lesions should not have received local treatment such as radiotherapy (lesions located within the previously treated area may also be targeted if progression is confirmed) .
4. ECOG physical strength score: 0-1;
5. Expected survival was ≥12 weeks;
6. 24-hour urine protein ≤1.0 g d) clotting: activated partial thromboplastin time (APTT) and international standard ratio (INR )≤1.5 × ULN (for use of a stable dose of anticoagulant therapy such as LMWH or Warfarin and INR can be screened within the expected range of anticoagulant therapy) ;
7. Eligible fertile patients (men and women) must agree to use a highly effective contraceptive method with their partner for at least 7 months during the trial and after the last dose; women of reproductive age must have a negative blood pregnancy test within 7 days before the first use of the study drug;
8. The subjects volunteered to join the study, signed the informed consent, good compliance, with follow-up.

Exclusion Criteria:

1. Subjects on systemic therapy with corticosteroid (> 10 mg daily equivalent of prednisone) or other immunosuppressive agents, except for local inflammation and the prevention of allergy and nausea and vomiting, who had undergone major surgery or severe trauma within 4 weeks prior to the first corticosteroid of the study drug, or who required elective surgery during the trial, who had undergone minor traumatic surgery, such as needle biopsy, within 7 days prior to the first dose of the study drug;
2. Previous allergies to monoclonal antibody, formulation components of SHR-A1811 products, and fluorouracil medications;
3. Previous antineoplastic therapy toxicities did not revert to a CTCAE v5.0 grade rating of ≤1(except for toxicities that the investigator judged to have no safety risk, such as alopecia, etc.) or the level specified by the enrollment/exclusion criteria;
4. Subjects with a history of meningeal metastasis or current meningeal metastasis; active brain metastasis;
5. uncontrolled pleural effusion, pericardial effusion, or ascites requiring repeated drainage;
6. history of immunodeficiency, these included people who tested positive for HIV or who had a fever of > 38.5 degrees of unknown cause before the first dose (cancer fever, as judged by the researchers, could be enrolled); Severe infection (CTCAE > Grade 2) occurred within 4 weeks before the first use of the study drug, such as severe pneumonia, bacteremia, infection complications, etc. Baseline chest imaging showed active pulmonary inflammation, active hepatitis B (HBV DNA ≥500 IU/mL) and hepatitis C (HCV-RNA was higher than the lower limit of detection);
7. Other malignancies in the past 5 years, not including cured skin basal-cell carcinoma and carcinoma in situ of the cervix;
8. Pregnant or lactating women.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Progressive free survive assessed by Independent Review Committee | Every 6 weeks, up to 3 years

SECONDARY OUTCOMES:
Security: adverse events | The first day of each cycle（21 days or 28 days）
Effectiveness: progressive free survive assessed by the researchers | Every 6 weeks, up to 3 years
Effectiveness: objective response rate assessed by the researchers | Every 6 weeks, up to 3 years
Effectiveness: duration of response assessed by the researchers | Every 6 weeks, up to 3 years
Effectiveness: overall survive assessed by the researchers | Every 6 weeks, up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided